CLINICAL TRIAL: NCT00679172
Title: A Randomised, Double-blind, Placebo-controlled, Single Dose, Dose Escalation Study to Determine the Immunogenicity, Safety and Tolerability of S. Typhi (Ty2 aroC-ssaV-) ZH9 at Doses of 5.0 x 10E9 CFU, 7.5 x 10E9 CFU, 1.1 x 10E10 and 1.7 x 10E10 CFU and 1.7 x 10E10 CFU, Following Oral Administration to Healthy, Typhoid Vaccine naïve Subjects in the USA.
Brief Title: Immunogenicity, Safety and Tolerability of the Typhoid Fever Vaccine Candidate M01ZH09 in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: MS01.13
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Typhoid
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- M01ZH09 Vaccine Candidate Cohort 1 (Experimental): Dose of 5.0 x 10^9 colony forming units (CFU) S. typhi (Ty2 aroC-ssaV-) ZH9 or placebo, administered as a single, oral dose
  Interventions: Biological: Dose of 5.0 x 10^9 CFU (Cohort 1); Other: Placebo (Cohorts 1-4 pooled)
- M01ZH09 Vaccine Candidate Cohort 2 (Experimental): Dose of 7.5 x 10^9 CFU S. typhi (Ty2 aroC-ssaV-) ZH9 or placebo, administered as a single, oral dose
  Interventions: Biological: Dose of 7.5 x 10^9 CFU (Cohort 2); Other: Placebo (Cohorts 1-4 pooled)
- M01ZH09 Vaccine Candidate Cohort 3 (Experimental): Dose of 1.1 x 10^10 CFU S. typhi (Ty2 aroC-ssaV-) ZH9 or placebo, administered as a single, oral dose
  Interventions: Biological: Dose of 1.1 x 10^10 CFU (Cohort 3); Other: Placebo (Cohorts 1-4 pooled)
- M01ZH09 Vaccine Candidate Cohort 4 (Experimental): Dose of of 1.7 x 10^10 CFU S. typhi (Ty2 aroC-ssaV-) ZH9 or placebo, administered as a single, oral dose
  Interventions: Biological: Dose of of 1.7 x 10^10 CFU (Cohort 4); Other: Placebo (Cohorts 1-4 pooled)

INTERVENTIONS:
Biological: Dose of 5.0 x 10^9 CFU (Cohort 1) — S. typhi (Ty2 aroC-ssaV-) ZH9 live attenuated typhoid vaccine, single dose, oral administration
  Arms: M01ZH09 Vaccine Candidate Cohort 1
Biological: Dose of 7.5 x 10^9 CFU (Cohort 2) — S. typhi (Ty2 aroC-ssaV-) ZH9 live attenuated typhoid vaccine, single dose, oral administration
  Arms: M01ZH09 Vaccine Candidate Cohort 2
Biological: Dose of 1.1 x 10^10 CFU (Cohort 3) — S. typhi (Ty2 aroC-ssaV-) ZH9 live attenuated typhoid vaccine, single dose, oral administration
  Arms: M01ZH09 Vaccine Candidate Cohort 3
Biological: Dose of of 1.7 x 10^10 CFU (Cohort 4) — S. typhi (Ty2 aroC-ssaV-) ZH9 live attenuated typhoid vaccine, single dose, oral administration
  Arms: M01ZH09 Vaccine Candidate Cohort 4
Other: Placebo (Cohorts 1-4 pooled) — Excipients only, single dose, oral administration

SUMMARY:
This study is to investigate the safety, tolerability and immunogenicity of the typhoid fever vaccine candidate M01ZH09 manufactured at commercial scale, at a new manufacturing facility. The vaccine will be delivered as a single oral dose to healthy, typhoid vaccine-naïve adults.

DETAILED DESCRIPTION:
This was a randomised, double-blind, placebo-controlled, single dose, dose escalation study with 4 dosing cohorts. Within each cohort, 45 evaluable subjects were planned (36 subjects receiving M01ZH09, 9 receiving placebo).

ELIGIBILITY:
Inclusion Criteria:

* healthy adult subjects aged 18 to 50 years inclusive, who are able and willing to give informed consent, following a detailed explanation of participation in protocol
* available for the duration of the study and available for scheduled and potential additional visits

Exclusion Criteria:

* women who are pregnant, breast-feeding or of childbearing potential and unwilling to use a reliable method of contraception throughout the study period
* history of anaphylactic shock following vaccination by any route have phenylketonuria
* hypersensitivity to any component of the vaccine or are hypersensitive to two of the following antibiotics: ciprofloxacin, azithromycin, ampicillin, trimethoprim sulfamethoxazole
* received antibiotic medication within 14 days prior to dosing
* received any vaccine within 4 weeks prior to dosing or plan to receive a vaccine within 4 weeks after dosing
* received any vaccine against Salmonella typhi (licensed or investigational) or ever suffered from typhoid fever
* subjects who test positive for hepatitis B, hepatitis C, HIV or human leucocyte antigen B-27
* known or suspected history of liver or active gall bladder disease, ongoing gastro-intestinal disease or abnormality
* commercial food handlers or health care workers with direct contact with high risk patients or who have household contacts with immuno-compromised individuals, pregnant women or children less than 2 years of age
* subjects who have a clinically significant amount of protein or haemoglobin in their urine or abnormality of their haematology or serum biochemistry parameters
* impairment of immune function or those receiving or have received cytotoxic drugs in the 6 months prior to study entry
* subjects who use antacids, proton pump inhibitors or H2 blockers on a regular basis or have consumed proton pump inhibitors or H2 blockers within 24 hours prior to dosing
* acute infections (including fever of 37.5 degrees Celsius or greater) on the day of dosing.
* subjects with chronic disease (e.g Crohn's disease, inflammatory bowel disease, diabetes) who cannot withstand a 3 hour fast
* substance abuse or a history of substance abuse that might interfere with participation in the study
* body mass index (BMI) is less than 19 or greater than 34 kg per m2
* clinically significant medical condition that precludes participation in the study
* subjects who have participated in an interventional clinical trial within 60 days of dosing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 187 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lockhart, DM, Study Director — Emergent BioSolutions
Locations (3):
- United States (3):
  - Miami Research Associates, South Miami, Florida
  - John Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - Unit of Infectious Diseases, University of Vermont College of Medicine, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lyon CE, Sadigh KS, Carmolli MP, Harro C, Sheldon E, Lindow JC, Larsson CJ, Martinez T, Feller A, Ventrone CH, Sack DA, DeNearing B, Fingar A, Pierce K, Dill EA, Schwartz HI, Beardsworth EE, Kilonzo B, May JP, Lam W, Upton A, Budhram R, Kirkpatrick BD. In a randomized, double-blinded, placebo-controlled trial, the single oral dose typhoid vaccine, M01ZH09, is safe and immunogenic at doses up to 1.7 x 10(10) colony-forming units. Vaccine. 2010 Apr 30;28(20):3602-8. doi: 10.1016/j.vaccine.2010.02.017. Epub 2010 Feb 24. PMID 20188175

RESULTS

PARTICIPANT FLOW:
Groups:
- M01ZH09 Vaccine Candidate Cohort 1: Dose of 5.0 x 10^9 CFU S. typhi (Ty2 aroC-ssaV-) ZH9.
- M01ZH09 Vaccine Candidate Cohort 2: Dose of 7.5 x 10^9 CFU S. typhi (Ty2 aroC-ssaV-) ZH9.
- M01ZH09 Vaccine Candidate Cohort 3: Dose of 1.1 x 10^10 CFU S. typhi (Ty2 aroC-ssaV-) ZH9.
- M01ZH09 Vaccine Candidate Cohort 4: Dose of 1.7 x 10^10 CFU S. typhi (Ty2 aroC-ssaV-) ZH9.
- Pooled Placebo: Placebo comparator comprised of excipients only, pooled across Cohorts 1-4.
Period: Overall Study
Arm/Group | M01ZH09 Vaccine Candidate Cohort 1 | M01ZH09 Vaccine Candidate Cohort 2 | M01ZH09 Vaccine Candidate Cohort 3 | M01ZH09 Vaccine Candidate Cohort 4 | Pooled Placebo
Started | 37 | 38 | 36 | 39 | 37
Completed | 36 | 37 | 35 | 38 | 37
Not Completed | 1 | 1 | 1 | 1 | 0
Not completed — Non-compliance | 1 | 1 | 0 | 1 | 0
Not completed — Other not specified | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | M01ZH09 Vaccine Candidate Cohort 1 | M01ZH09 Vaccine Candidate Cohort 2 | M01ZH09 Vaccine Candidate Cohort 3 | M01ZH09 Vaccine Candidate Cohort 4 | Pooled Placebo | Total
Number analyzed (Participants) | 37 | 38 | 36 | 39 | 37 | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1 | 1 | 1 | 4
  Between 18 and 65 years | 36 | 38 | 35 | 38 | 36 | 183
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (10.13) | 33.1 (10.00) | 32.0 (9.99) | 31.3 (9.21) | 32.3 (10.01) | 32.4 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 19 | 19 | 21 | 94
  Male | 19 | 21 | 17 | 20 | 16 | 93
Region of Enrollment [Number; unit: participants]
  United States | 37 | 38 | 36 | 39 | 37 | 187

OUTCOME MEASURES:

1. Primary Outcome: Number and Proportion of Subjects Reporting Suspected Unexpected Serious Adverse Reactions.
Description: Number and proportion of subjects reporting suspected unexpected serious adverse reactions (SUSARs).
Time Frame: From start of dosing to 28 days post-dosing.
Population: Safety Population: All subjects who received a dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | M01ZH09 Vaccine Candidate Cohort 1 | M01ZH09 Vaccine Candidate Cohort 2 | M01ZH09 Vaccine Candidate Cohort 3 | M01ZH09 Vaccine Candidate Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 37 | 38 | 36 | 39 | 37
Participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number and Proportion of Subjects Experiencing Symptomatic Fever.
Description: Number and proportion of subjects experiencing symptomatic (e.g., chills, rigors, sweating, headache, myalgia etc.) elevated body temperature of 38.0°C or more in the 14 days following dosing.
Time Frame: From start of dosing to 14 days post-dosing.
Population: Safety Population: All subjects who received a dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | M01ZH09 Vaccine Candidate Cohort 1 | M01ZH09 Vaccine Candidate Cohort 2 | M01ZH09 Vaccine Candidate Cohort 3 | M01ZH09 Vaccine Candidate Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 37 | 38 | 36 | 39 | 37
Participants | 1 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Subjects Having Clinically Significant Changes in Laboratory Test Parameters.
Description: Number of subjects having clinically significant changes in clinical laboratory test parameters.
Time Frame: From start of dosing to 28 days post-dosing.
Population: Safety Population: All subjects who received a dose of study medication.
Measure: Number; unit: participants
Arm/Group | M01ZH09 Vaccine Candidate Cohort 1 | M01ZH09 Vaccine Candidate Cohort 2 | M01ZH09 Vaccine Candidate Cohort 3 | M01ZH09 Vaccine Candidate Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 37 | 38 | 36 | 39 | 37
participants
  Alanine aminotransferase | 1 | 0 | 0 | 0 | 0
  Creatinine | 0 | 0 | 0 | 0 | 0
  Eosinophils | 0 | 0 | 0 | 0 | 0
  Haematocrit | 0 | 0 | 0 | 1 | 0
  Haemoglobin | 0 | 0 | 0 | 1 | 0
  Lymphocytes | 0 | 0 | 0 | 0 | 1
  Neutrophils | 0 | 0 | 0 | 0 | 1
  Platelet Count | 0 | 0 | 0 | 0 | 0
  Red Blood Cell Count | 0 | 0 | 0 | 1 | 0
  White Blood Cell Count | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Subjects Reporting Treatment-related TEAEs.
Description: Number of subjects having TEAEs considered by the principal investigator to be "possibly" or "probably" related to treatment.
Time Frame: From start of dosing to 28 days post-dosing.
Population: Safety Population: All subjects who received a dose of study medication.
Measure: Number; unit: participants
Arm/Group | M01ZH09 Vaccine Candidate Cohort 1 | M01ZH09 Vaccine Candidate Cohort 2 | M01ZH09 Vaccine Candidate Cohort 3 | M01ZH09 Vaccine Candidate Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 37 | 38 | 36 | 39 | 37
participants
  Subjects with possibly related TEAEs | 19 | 12 | 18 | 10 | 15
  Subjects with probably related TEAEs | 7 | 10 | 6 | 19 | 9

5. Primary Outcome: Number and Proportion of Subjects Experiencing Bacteraemia.
Description: Number and proportion of subjects experiencing a proven bacteraemia attributed to the vaccine strain S. typhi (Ty2 aroC-ssaV-) ZH9.
Time Frame: From start of dosing to 28 days post-dosing.
Population: Safety Population: All subjects who received a dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | M01ZH09 Vaccine Candidate Cohort 1 | M01ZH09 Vaccine Candidate Cohort 2 | M01ZH09 Vaccine Candidate Cohort 3 | M01ZH09 Vaccine Candidate Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 37 | 38 | 36 | 39 | 37
Participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Subjects Having Shedding in Stool of Salmonella Typhi (S. Typhi) (Ty2 aroC-ssaV-) ZH9.
Description: Number of subjects having shedding in stool of S. typhi (Ty2 aroC-ssaV-) ZH9. Subjects were evaluated beyond Day 14 only in Cohort 4.
Time Frame: Beyond 7 days post-dosing through 14 days post-dosing (Cohorts 1-3) or through 21 days post-dosing (Cohort 4).
Population: Safety Population: All subjects who received a dose of study medication.
Measure: Number; unit: participants
Arm/Group | M01ZH09 Vaccine Candidate Cohort 1 | M01ZH09 Vaccine Candidate Cohort 2 | M01ZH09 Vaccine Candidate Cohort 3 | M01ZH09 Vaccine Candidate Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 37 | 38 | 36 | 39 | 37
participants
  Day 9: number analyzed (Participants) | 35 | 35 | 34 | 38 | 37
  Day 9 | 1 | 0 | 1 | 1 | 0
  Day 11: number analyzed (Participants) | 34 | 36 | 35 | 36 | 34
  Day 11 | 0 | 1 | 0 | 2 | 0
  Day 14: number analyzed (Participants) | 36 | 37 | 36 | 37 | 35
  Day 14 | 0 | 0 | 0 | 1 | 0
  Day 17: number analyzed (Participants) | 0 | 0 | 0 | 37 | 9
  Day 17 |  |  |  | 2 | 0
  Day 19: number analyzed (Participants) | 0 | 0 | 0 | 34 | 9
  Day 19 |  |  |  | 0 | 0
  Day 21: number analyzed (Participants) | 0 | 0 | 0 | 37 | 9
  Day 21 |  |  |  | 0 | 0

7. Primary Outcome: Number and Proportion of Subjects Developing an Immune Response as Determined by the Level of IgG and/or IgA Antibodies for S. Typhi Lipopolysaccharide (LPS).
Description: Number and proportion of subjects with increase of 70% (fold change of 1.7) in S. typhi LPS-specific serum IgG at Days 14 or 28 AND/OR increase of 50% (fold change of 1.5) in S. typhi LPS-specific serum IgA at Days 7 or 14. Serum IgG and IgA were assayed using enzyme-linked immunosorbent assay (ELISA).
Time Frame: From baseline (pre-dose) to Days 14 or 28 (IgG) or to Days 7 or 14 (IgA).
Population: ITT Population: all subjects who received study medication and had any postbaseline immunogenicity data available up to and including Day 28.
Measure: Count of Participants; unit: Participants
Groups:
- M01ZH09 Vaccine Candidate Cohort 4: Dose of 1.7 x 10^10 CFU S. typhi (Ty2 aroC- ssaV-) ZH9.
Arm/Group | M01ZH09 Vaccine Candidate Cohort 1 | M01ZH09 Vaccine Candidate Cohort 2 | M01ZH09 Vaccine Candidate Cohort 3 | M01ZH09 Vaccine Candidate Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 37 | 38 | 36 | 39 | 37
Participants | 32 | 35 | 32 | 38 | 6

8. Secondary Outcome: Number and Proportion of Subjects Developing an Immune Response as Determined by the Level of IgA Antibodies for S. Typhi LPS.
Description: Number and proportion of subjects with increase of 50% (fold change of 1.5) in S. typhi LPS-specific serum IgA at Days 7 or 14. Serum IgA was assayed using ELISA.
Time Frame: From baseline (pre-dose) to Days 7 or 14.
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | M01ZH09 Vaccine Candidate Cohort 1 | M01ZH09 Vaccine Candidate Cohort 2 | M01ZH09 Vaccine Candidate Cohort 3 | M01ZH09 Vaccine Candidate Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 37 | 38 | 36 | 39 | 37
Participants | 31 | 35 | 30 | 38 | 1

9. Secondary Outcome: Number and Proportion of Subjects Developing an Immune Response as Determined by the Level of IgG Antibodies for S. Typhi LPS.
Description: Number and proportion of subjects with increase of 70% (fold change of 1.7) in S. typhi LPS-specific serum IgG at Days 14 or 28. Serum IgG was assayed using ELISA.
Time Frame: From baseline (pre-dose) to Days 14 or 28.
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | M01ZH09 Vaccine Candidate Cohort 1 | M01ZH09 Vaccine Candidate Cohort 2 | M01ZH09 Vaccine Candidate Cohort 3 | M01ZH09 Vaccine Candidate Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 37 | 38 | 36 | 39 | 37
Participants | 23 | 30 | 31 | 33 | 5

10. Secondary Outcome: Number and Proportion of Subjects Developing an Immune Response as Determined by the Level of IgG Antibodies for S. Typhi LPS.
Description: Number and proportion of subjects with an increase of 70% (fold change of 1.7) in S. typhi LPS-specific serum IgG at Days 7, 14 or 28. Serum IgG was assayed using ELISA.
Time Frame: From baseline (pre-dose) to Days 7, 14, or 28.
Population: ITT Population: all subjects who received study medication and had any postbaseline immunogenicity data available up to and including Day 14.
Measure: Count of Participants; unit: Participants
Arm/Group | M01ZH09 Vaccine Candidate Cohort 1 | M01ZH09 Vaccine Candidate Cohort 2 | M01ZH09 Vaccine Candidate Cohort 3 | M01ZH09 Vaccine Candidate Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 37 | 38 | 36 | 39 | 37
Participants | 25 | 30 | 31 | 33 | 7

11. Secondary Outcome: Number and Proportion of Subjects Developing an Immune Response at the Target Dose of 7.5 x 10^9 CFU (Cohort 2) as Determined by the Number of Antibody Secreting Cells (ASCs) Secreting IgA and/or Fold Change in IgG.
Description: Number and proportion of subjects with ≥ 4 ASCs per 10^6 peripheral blood mononuclear cells (PBMCs) at Day 7 secreting IgA specific for S. typhi LPS (detected by enzyme-linked immunospot assay [ELISPOT]) AND/OR 4-fold increase for serum IgG on Day 28 compared to baseline (assay using endpoint titre ELISA).
Time Frame: At Day 7 (IgA); and from baseline (pre-dose) to Day 28 (IgG).
Population: ITT Population (Cohort 2): all subjects who received study medication and had any postbaseline immunogenicity data available up to and including Day 28.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo - Cohort 2: Placebo comparator comprised of excipients only - Cohort 2
Arm/Group | M01ZH09 Vaccine Candidate Cohort 2 | Placebo - Cohort 2
Number analyzed (Participants) | 38 | 9
Participants | 36 | 0

12. Secondary Outcome: Number and Proportion of Subjects Developing an Immune Response at the Target Dose of 7.5 x 10^9 CFU (Cohort 2) as Determined by the Number of ASCs Secreting IgA.
Description: Number and proportion of subjects with ≥ 4 ASCs per 10^6 PBMCs at Day 7 secreting IgA specific for S. typhi LPS (detected by ELISPOT).
Time Frame: Day 7.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | M01ZH09 Vaccine Candidate Cohort 2 | Placebo - Cohort 2
Number analyzed (Participants) | 38 | 9
Participants | 35 | 0

13. Secondary Outcome: Number and Proportion of Subjects Developing an Immune Response at the Target Dose of 7.5 x 10^9 CFU (Cohort 2) as Determined by the Fold Change in IgG.
Description: Number and proportion of subjects with 4-fold increase for serum IgG on Day 28 compared to baseline (assay using endpoint titre ELISA).
Time Frame: From baseline (pre-dose) to Day 28.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | M01ZH09 Vaccine Candidate Cohort 2 | Placebo - Cohort 2
Number analyzed (Participants) | 38 | 9
Participants | 14 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 28.
Description: Treatment-emergent adverse events (TEAEs) are defined as those adverse events which occurred postdose or which were present predose and became worse postdose. The proportions of subjects reported TEAEs and SAEs were pre-defined safety outcome variables.
Arm/Group | M01ZH09 Vaccine Candidate Cohort 1 | M01ZH09 Vaccine Candidate Cohort 2 | M01ZH09 Vaccine Candidate Cohort 3 | M01ZH09 Vaccine Candidate Cohort 4 | Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38 | 0/36 | 0/39 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38 | 0/36 | 0/39 | 0/37
Other Adverse Events (participants affected / at risk) | 27/37 | 26/38 | 30/36 | 33/39 | 31/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | M01ZH09 Vaccine Candidate Cohort 1 (N=37) | M01ZH09 Vaccine Candidate Cohort 2 (N=38) | M01ZH09 Vaccine Candidate Cohort 3 (N=36) | M01ZH09 Vaccine Candidate Cohort 4 (N=39) | Pooled Placebo (N=37)
Abdominal pain (Gastrointestinal disorders) | 11 | 12 | 7 | 12 | 8
Constipation (Gastrointestinal disorders) | 7 | 4 | 1 | 5 | 8
Diarrhoea (Gastrointestinal disorders) | 5 | 10 | 6 | 9 | 10
Flatulence (Gastrointestinal disorders) | 17 | 15 | 10 | 10 | 14
Nausea (Gastrointestinal disorders) | 9 | 6 | 3 | 10 | 5
Asthenia (General disorders) | 8 | 13 | 6 | 7 | 8
Anorexia (Metabolism and nutrition disorders) | 3 | 8 | 1 | 4 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 6 | 3 | 7 | 7
Headache (Nervous system disorders) | 16 | 5 | 9 | 15 | 13
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0
Chills (General disorders) | 2 | 0 | 2 | 7 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 4 | 3
Culture stool positive (Investigations) | 1 | 1 | 1 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0/18 | 1/17 | 2/19 | 1/19 | 1/21
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any proposed publication was subject to review conditions and timelines agreed between Emergent Product Development UK Ltd and the site Principal Investigator and detailed in the agreements with these parties prior to the start of the study.